CLINICAL TRIAL: NCT02627222
Title: The Efficacy of Pro-vitamin A Biofortified Cassava on Vitamin A Status in Nigerian Preschool Children
Acronym: CASSAVITA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: University of Ibadan (Other); International Institute for Tropical Agriculture (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CASSAVITA II
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Vitamin A Deficiency
Keywords: Pro-vitamin A; Cassava; Vitamin A deficiency; Retinol Isotope Dilution; Preschool children; Nigeria
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Daily consumption of two cassava-based meals prepared with pro-vitamin A rich biofortified cassava
  Interventions: Other: Pro-vitamin A biofortified cassava
- Control (Placebo Comparator): Daily consumption of two cassava-based meals prepared with common white cassava
  Interventions: Other: White cassava

INTERVENTIONS:
Other: Pro-vitamin A biofortified cassava — Pro-vitamin A biofortified cassava is the product of international conventional breeding programs (non-GMO) in order to increase the pro-vitamin A content of cassava for improved nutritional intake
  Other Names: Yellow cassava; Biofortified cassava
  Arms: Treatment
Other: White cassava — Conventional white cassava
  Other Names: Cassava; Manihot esculenta
  Arms: Control

SUMMARY:
The study comprises an open-label randomized controlled trial investigating the efficacy of consuming a daily ration of pro-vitamin A biofortified cassava on vitamin A status of Nigerian children, aged 3-4 years old (n=200).

DETAILED DESCRIPTION:
Objective: The primary objective is to assess the efficacy of daily consumption of pro-vitamin A rich cassava during 10 weeks on body retinol pools of 3-4 year old children in Nigeria after high-dose vitamin A supplementation. The secondary objectives are: 1) To investigate the effect of daily consumption of pro-vitamin A rich cassava on functional indicators such as nutritional anaemia and gut integrity; 2) To investigate the effect of zinc deficiency and genetic polymorphisms in the Beta-Carotene Oxygenase 1 (BCO1) and related genes on the efficacy of pro-vitamin A rich cassava consumption; 3) To compare the skin colour in the palm of the hand of each participant with their serum retinol levels using a handheld non-invasive spectrophotometer.

Study design: Open-label (single-blinded) randomized controlled trial with two parallel groups Study population: Pre-school children, aged 3-4 years living in Osun State area, South-Western Nigeria. Children (n=750) will be screened for eligibility. Out of these, n=250 will undergo a 4-week run-in phase. n=200 children will be randomly allocated to two different treatments: 1) Yellow cassava providing ~50% of the recommended daily allowance (RDA) for vitamin A; 2) White cassava.

Main study parameters/endpoints: The primary outcome was the difference in body retinol pools between groups 1 and 2 at the end of intervention; however, due to the inability to assess body retinol pools, the modified primary outcome is the difference in serum retinol concentrations between groups 1 and 2. Other outcome measures include: other vitamin A status indicators (β-carotene, retinol binding protein, transthyretin), inflammatory markers, iron status indicators, anthropometrics, gut integrity, and thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 36 - 59 months (verified by birth certificates, vaccination cards or other formal documentation)
* Apparently healthy
* Parental informed consent

Exclusion Criteria:

* Frequently absent (>20% of feeding days) during run-in
* Children not assenting during blood collections
* Signs or history of infectious or systemic diseases (e.g. tuberculosis, sickle cell anaemia)
* Mental status that is incompatible with the proper conduct of the study
* Current participation in other research
* Food allergy related to the intervention foods

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Body retinol pool (omitted) | 13 weeks
  Difference in body retinol pools between groups
(Modified primary outcome): Serum retinol | 13 weeks
  Difference in serum retinol pools between groups

SECONDARY OUTCOMES:
Anaemia | 13 weeks
  Difference in haemoglobin concentration between groups
Gut integrity | 11 weeks
  Difference in gut integrity between groups

OTHER OUTCOMES:
Serum betacarotene | 13 weeks
  Difference in serum retinol concentration between groups
Retinol binding protein | 13 weeks
  Difference in serum retinol binding protein concentration between groups
Urinary thiocyanate | 11 weeks
  Difference in urinary thiocyanate concentration between groups
Thyroid function indicators | 13 weeks
  Difference in serum thyroid function indicators between groups
Serum zinc | Baseline
  Effect modification by baseline zinc deficiency
Genetic polymorphisms in the BCO1 gene | Baseline
  Effect modification by BCO1 polymorphisms
Inflammatory markers | Baseline and end of study
  C-reactive protein, alpha glycoprotein
Malaria | Baseline and end of study
  A-symptomatic malaria

CONTACTS AND LOCATIONS:
Overall Officials: Alida Melse-Boonstra, PhD, Principal Investigator — Division of Human Nutrition, Wageningen University
Locations (1):
- Department of Human Nutrition, University of Ibadan, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Afolami I, Mwangi MN, Samuel F, Boy E, Ilona P, Talsma EF, Feskens E, Melse-Boonstra A. Daily consumption of pro-vitamin A biofortified (yellow) cassava improves serum retinol concentrations in preschool children in Nigeria: a randomized controlled trial. Am J Clin Nutr. 2021 Jan 4;113(1):221-231. doi: 10.1093/ajcn/nqaa290. PMID 33184647